CLINICAL TRIAL: NCT03781531
Title: Identification of Novel Biomarkers to Aid in the Detection of Occult Cancer in Patients With Venous Thromboembolism
Status: Recruiting | Type: Observational
Sponsor: Danderyd Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: dnr2017/260-31/4
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Cancer; Venous Thromboembolism
Keywords: Occult cancer; Venous thromboembolism; Biomarkers; Early diagnosis; Neutrophil extracellular traps
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Venous thromboembolism: Patients presenting with venous thromboembolism (thrombosis in the deep venous system of upper or lower extremities or iliac veins and/or pulmonary embolism) as detected by ultrasonography, phlebography, computer tomography, or angiography

SUMMARY:
Venous thromboembolism is a common and serious complication in cancer, and is associated with a substantially increased morbidity and mortality. Furthermore, VTE may be the earliest sign of cancer. Recent studies, however, fail to show a clinical benefit of extended cancer screening in this patient population. Better risk prediction models are therefore warranted to identify VTE patients who would benefit from a rapid and extensive cancer screening. Inflammation and hypercoagulability are considered hallmarks of cancer, and emerging light is being shed on the potential of various markers of inflammation and coagulation in cancer diagnostics and prognostics. Among the inflammatory and thrombotic processes linked to cancer is the neutrophil release of web-like nuclear chromatin (DNA and histones), referred to as neutrophil extracellular traps (NETs). Driven by the tumor environment, NETs have recently been shown to play a central role in tumor progression, metastasis, and tumor-associated thrombosis.

The investigators hypothesize that an enhanced inflammatory state may be predictive of an underlying cancer in patients presenting with VTE. The present study is an ongoing prospective study with the primary aim to investigate the diagnostic potential of markers of inflammation, including markers of NETs, in detecting occult cancer in patients presenting with VTE. Secondary aims are to include other biomarkers of cancer, and to assess whether any or a combination of these biomarkers may be prognostic of occult cancer, recurrent thrombotic events, mortality, or cancer disease progression in VTE patients with an underlying malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Venous thromboembolism (thrombosis in the deep venous system of upper or lower extremities or iliac veins and/or pulmonary embolism) as detected by ultrasonography, phlebography, computer tomography, or angiography;
* > 18 years or older;
* Written informed consent

Exclusion Criteria:

* > 2 days after VTE diagnosis;
* No blood withdrawal at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients age >18 years with objectively confirmed venous thromboembolism (thrombosis in the deep venous system of upper or lower extremities or iliac veins and/or pulmonary embolism) diagnosed < 2 days.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cancer | Within 2 years from study inclusion
  Patients diagnosed with VTE will be referred for a limited cancer screening according to current guidelines. Cancer diagnosis - if not present at inclusion - will be obtained during a two-year follow-up from hospital records and/or the Swedish cancer registry

SECONDARY OUTCOMES:
Recurrent thrombotic event | Within 2 years from study inclusion
  Recurrent thrombotic event (arterial or venous thrombosis) will be obtained during a two-year follow-up from hospital records and/or the Swedish national patient registry
All-cause mortality | Within 2 years from study inclusion
  All-cause mortality will be obtained during a two-year follow-up from hospital records and/or the Swedish death registry
Cancer progression among enrolled patients with a cancer diagnosis at study inclusion | Within 2 years from study inclusion
  Patients with cancer progression will be identified during a two-year follow-up from hospital records and/or the Swedish cancer registry

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Thålin, M.D., Ph.D., Principal Investigator — Karolinska Institutet; Håkan Wallén, M.D., Prof., Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Danderyd Hospital, Stockholm
  - Södersjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided